CLINICAL TRIAL: NCT04424394
Title: A Pilot Study to Evaluate the Immediate and Short-term Efficacy of DualStim (Focused and Radial Extracorporeal Shock Wave) Therapy With and Without Intracavernosal Wharton's Jelly in Patients With Erectile Dysfunction
Brief Title: DualStim Therapy With or Without Umbilical Cord Derived Wharton's Jelly for Erectile Dysfunction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BioIntegrate (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOINT - 2020DSWJ/ED
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- DualStim Therapy with Wharton's Jelly Injection (Experimental): DualStim therapy with intracavernosal injection of umbilical cord-derived Wharton's Jelly formulation.
  Interventions: Device: DualStim Therapy; Biological: Umbilical cord-derived Wharton's Jelly
- DualStim Therapy without Wharton's Jelly Injection (Active Comparator): DualStim therapy with intracavernosal injection of normal saline.
  Interventions: Device: DualStim Therapy; Other: Saline

INTERVENTIONS:
Device: DualStim Therapy — 6 DualStim Therapies over a period of 7 weeks.
Biological: Umbilical cord-derived Wharton's Jelly — 2 intracavernosal injections over a period of 7 weeks.
  Arms: DualStim Therapy with Wharton's Jelly Injection
Other: Saline — 2 intracavernosal injections over a period of 7 weeks.
  Arms: DualStim Therapy without Wharton's Jelly Injection

SUMMARY:
The purpose of this study is to determine the immediate and short-term efficacy of the methodological application of DualStim Therapy - Focused Extracorporeal Shock Wave Therapy (fESWT) and Radial Extracorporeal Shock Wave Therapy (rESWT), with and without intracavernosal administration of formulated umbilical cord derived Wharton's Jelly to improve and/or restore erectile function in patients with erectile dysfunction (ED).

DETAILED DESCRIPTION:
Erectile Dysfunction (ED) is broadly defined as the inability to achieve or maintain an erection sufficient for sexual intercourse or activity. Current treatment for ED consists of oral medications, vacuum devices, intracavernosal injections, and surgically placed penile prosthetics. In the literature, this has been described as a Stepwise Approach, offering therapy beginning with the least invasive treatment option.

The low intensity extracorporeal shock wave therapy (LISWT) was recently approved by the FDA for treatment of diabetic ulcers. But it is still under evaluation for treatment of ED. Recently, the European Association of Urology updated their guidelines related to ED and included LISWT for men with mild to moderate ED. Studies have reported that LISWT can be effective in treating ED. This was attributed to increase in angiogenesis, neurogenesis and other rejuvenating tissue effects. Doppler ultrasound studies have demonstrated a sustained increase in blood flow in patients treated with LISWT. Published studies have also reported a response rate of 40-80% with this treatment. In addition, the energy/pulse used in this application is approximately 10% of the energy used for disintegrating kidney stones; and no serious side effects have been reported till date.

Additionally, most completed studies included men who score in the moderate to minimal ranges on the International Index of Erectile Function. In the proposed study, men with severe to moderate ED based on IIEF-EF score will be included. The goal of this study is to improve and/or restore erectile function in men with erectile dysfunction. The investigators hypothesize (Alternate Hypothesis) that patients in the active treatment group (DualStim + Wharton's Jelly) will show an improvement of at least 4 points for moderate ED and at least 7 points for severe ED on IIEF-EF scale/questionnaire, and this difference will be significantly different from their baseline. In addition, patients in the DualStim + Saline group will be significantly different from their baseline, however, will show less improvement compared to DualStim + Wharton's Jelly. Our null hypothesis is that there is no difference between DualStim with Saline and DualStim with Wharton's Jelly groups and no difference between the baseline and after-treatment within the treatment groups for alleviating ED measured using International Index of Erectile Function score (IIEF-EF).

ELIGIBILITY:
Inclusion Criteria:

1. Only Male patients who are 40 to 80 years old (both numbers inclusive).
2. Must have a body mass index (BMI) of less than 35.
3. Patients with ED for at least 1 year but less than 10 years.
4. The patient is poorly phosphodiesterase type 5 inhibitors responsive, meaning he is able to achieve an erection but is unable or partially able to satisfactory complete sexual intercourse (penetration and/or orgasm).
5. Minimum IIEF-EF domain score of 11-16 (for classification as moderate ED).
6. IIEF-ED score ≥11 and ≤25 while taking phosphodiesterase type 5 inhibitors or in injection therapy.
7. Be willing and capable of giving written informed consent to participate in this clinical study.
8. Be willing and capable of complying with study-related requirements, procedures and visits.

Exclusion Criteria:

1. Patients with history of radical prostatectomy or extensive pelvic surgery.
2. Patients with past radiation therapy of the pelvic region within 12 months prior to enrollment.
3. Patients recovering from cancer within 12 months prior to enrollment.
4. Patients who are taking blood thinners or have history of Diabetes Mellitus.
5. Patients with untreated hypogonadism or thyroid disease.
6. Patients with deformed Penis on physical exam form.
7. Patients who participated in another clinical trial or treatment with any investigational product within last 30 days prior to inclusion in the study.
8. Patients with serious neurological, psychological or psychiatric disorders which may affect erectile function.
9. Patients with other medical conditions determined by site principal investigator as interfering with the study.
10. Patients with an injury or disability claim under current litigation or pending or approved workers' compensation claim.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only Male patients are eligible to participate.
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse or Severe adverse events associated with Intracavernosal administration of umbilical cord derived Wharton's Jelly injection. | During the procedure
  To determine the safety i.e. adverse or severe adverse events associated with intracavernosal administration of umbilical cord derived Wharton's Jelly injection. Any adverse or severe adverse events will be recorded in the associated case report forms.
Adverse or Severe adverse events associated with Intracavernosal administration of umbilical cord derived Wharton's Jelly injection. | 1 month follow-up visit
  To determine the safety i.e. adverse or severe adverse events associated with intracavernosal administration of umbilical cord derived Wharton's Jelly injection. Any adverse or severe adverse events will be recorded in the associated case report forms.
Adverse or Severe adverse events associated with Intracavernosal administration of umbilical cord derived Wharton's Jelly injection. | 3 month follow-up visit
  To determine the safety i.e. adverse or severe adverse events associated with intracavernosal administration of umbilical cord derived Wharton's Jelly injection. Any adverse or severe adverse events will be recorded in the associated case report forms.
Adverse or Severe adverse events associated with Intracavernosal administration of umbilical cord derived Wharton's Jelly injection. | 6 month follow-up visit
  To determine the safety i.e. adverse or severe adverse events associated with intracavernosal administration of umbilical cord derived Wharton's Jelly injection. Any adverse or severe adverse events will be recorded in the associated case report forms.
Adverse or Severe adverse events associated with Intracavernosal administration of umbilical cord derived Wharton's Jelly injection. | 12 month follow-up visit
  To determine the safety i.e. adverse or severe adverse events associated with intracavernosal administration of umbilical cord derived Wharton's Jelly injection. Any adverse or severe adverse events will be recorded in the associated case report forms.
Adverse or Severe adverse events associated with Intracavernosal administration of umbilical cord derived Wharton's Jelly injection. | 18 month follow-up visit
  To determine the safety i.e. adverse or severe adverse events associated with intracavernosal administration of umbilical cord derived Wharton's Jelly injection. Any adverse or severe adverse events will be recorded in the associated case report forms.
Immediate and short-term efficacy of DualStim Therapy with Wharton's Jelly based on changes in the International Index of Erectile Function Questionnaire score compared to baseline | through study completion, an average of 18 months
  To evaluate the immediate and short-term efficacy of DualStim Therapy with Wharton's Jelly based on changes in the International Index of Erectile Function Questionnaire score compared to baseline score. An increase in the score indicates improvement.

SECONDARY OUTCOMES:
Immediate and short-term efficacy of DualStim Therapy with Wharton's Jelly compared to DualStim Therapy with saline based on changes in the International Index of Erectile Function Questionnaire score. | through study completion, an average of 18 months
  To evaluate the immediate and short-term efficacy of DualStim Therapy with Wharton's Jelly compared to DualStim Therapy with saline based on changes in the International Index of Erectile Function Questionnaire score at each time-point.
Sexual activity improvement according to Sexual Encounter Profile Questionnaire from baseline leading to optimal penetration at follow-ups | through study completion, an average of 18 months
  To study sexual activity improvement from baseline leading to optimal penetration at follow-ups 1, 3 and 6 months' post treatment according to Sexual Encounter Profile Questionnaire. An increase in score indicates improvement.
Sexual activity improvement according to Global Assessment Questionnaire from baseline leading to optimal penetration at follow-ups | through study completion, an average of 18 months
  To study sexual activity improvement from baseline leading to optimal penetration at follow-ups 1, 3 and 6 months' post treatment according to Global Assessment Questionnaire. An increase in score indicates improvement.
Sexual activity improvement according to Erection Hardness Score from baseline leading to optimal penetration at follow-ups | through study completion, an average of 18 months
  To study sexual activity improvement from baseline leading to optimal penetration at follow-ups 1, 3 and 6 months' post treatment according to Erection Hardness Score. An increase in score indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gaines, MD, Principal Investigator — LifeGAINES Medical and Aesthetics Center; Ashim Gupta, PhD, MBA, Study Director — BioIntegrate

IPD SHARING:
Plan to Share IPD: No